CLINICAL TRIAL: NCT04978792
Title: Does Cultivating Self-compassion Improve Resilience to Criticism and Improve Mental Health in Adults With ADHD?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Principal Investigator, Danielle Beaton, Principle Investigator, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 172839
Record Dates: First submitted 2021-07-09; First posted 2021-07-27 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: ADHD; Depression; Stress; Self-Criticism; Anxiety; Wellbeing; Self-compassion
Keywords: self-compassion; criticism; ADHD; mental health
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-compassion Intervention (Experimental): The intervention will include 14 self-compassion exercises completed over a 3-week period. The intervention will include methods of psychoeducation, meditation, and self-compassion exercises similar to Beshai et al.'s (2020) self-compassion-based intervention. The psychoeducation will focus on self-compassion, the meditations will be kindness and loving meditations and self-compassion breaks. The self-compassion exercises will be based on the writing exercises available on Neff's self-compassion website.
  Interventions: Behavioral: Online self-compassion intervention
- Control Group (Active Comparator): The active control will also include 14 exercises completed over a 3-week period. The 14 exercises will comprise of a psychoeducation video, writing exercises, video/audio-guided relaxation, and journal entries. The same psychoeducation video used in the intervention will be shown to participants, however, the other exercises will be altered to focus on factual information and not focused on self-compassion. The exercises will be matched to the self-compassion exercise so that similar exercises are completed in parallel time with the intervention.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Online self-compassion intervention — An online self-guided intervention that uses widely available exercises and information.
  Arms: Self-compassion Intervention
Behavioral: Active Control — Participants will complete written exercises and breathing exercises that are not associated with self-compassion
  Arms: Control Group

SUMMARY:
This study aims to investigate the effect that increasing levels of self-compassion may have on levels of perceived criticism, self-criticism, and mental health of adults with ADHD. A secondary aim of the study is to capture how feasible using an online self-guided self-compassion practice maybe with people with ADHD.

Research Questions

1. Does a short self-guided self-compassion intervention increase levels of state and/or trait self-compassion in adults with ADHD over time?
2. Are changes in state and/or trait self-compassion associated with changes in levels of self-criticism or perceived criticism?
3. Are changes in state and/or trait self-compassion associated with improvements in mental health?
4. Are changes in mental health mediated by changes in self-criticism or perceived criticism?

ELIGIBILITY:
Inclusion Criteria:

* Self-report a formal diagnosis of ADHD
* Scores on the Adult ADHD Self Report Questionnaire (ASRS) meet the clinical cut-off.
* No previous engagement with self-compassion interventions/practice

Exclusion Criteria:

* No previous experiences of trauma.
* No PTSD
* No personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in trait Self-compassion | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The self-compassion scale (SCS, Neff, 2003) consists of 26 items measured on a scale between 1-5 (never - always). The items include 3 sub-scales that represent compassionate self-responding (self-kindness, mindfulness and common humanity) and 3 sub-scales of uncompassionate self-responding (self-judgement, isolation and over-identification). To obtain a total self-compassion score, the uncompassionate items are reverse coded, the mean score for each subscale is calculated, then the mean of the six subscale scores added together is calculated. The mean scores can range between 1 - 5, whereby higher scores indicate higher self-compassion
Change in state self-compassion | 4x a week after intervention exercise complete.
  The State Self-Compassion Scale Short Form (SSCS-S; (Neff et al., 2021) is a six-item measure of state self-compassion. The six items are rated on a 5-point scale from 1 (not at all true for me) to 5 (very true for me), and responses are summed (after negatively worded questions are reverse coded) to provide a global state self-compassion measure. Higher scores equate to higher levels of state self-compassion.
Change in Perceived Criticism | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  An adapted version of The Perceived Criticism Scale (PCS) (Hooley & Teasdale, 1989) will be used to measure how much criticism is "getting through" to individuals. The measure is a single question, "How critical do you think people in your nearest environment - such as family, friends, colleagues - are of you?", that is rated between 0 (not at all critical of me) to 10 (very critical of me). The measure can also include a second item also rated on a 1-10 scale that asks how upset the respondent may become when criticised.
Change in wellbeing | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The Mental Health Continuum Short Form (MHC-SF) (Keyes, 2009) will be used to measure the frequency of well-being symptoms (never [0] - every day [5]). The self-report questionnaire includes 14-items that measure emotional well-being (3-items), psychological well-being (6-items) and social well-being (5-items). A global well-being score between 0 - 70 is achieved by summing the scores for each item, whereby higher scores equal greater well-being. Subscale scores are calculated by summing the responses for each item of the corresponding sub-scale; emotional well-being scores can range between 0 - 15, social well-being scores can range between 0 - 25, and psychological well-being scores can range between 0 - 30.
Change in Depression | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The Patient Health Questionnaire - 9 (PHQ-9) (Kroenke et al., 2001) will be used to assess the severity of depressive symptoms and assess responses to treatment. The PHQ-9 has nine items that represent each of the DSM-IV (APA) criteria of depression. The items, such as "feeling down, depressed, or hopeless?", are rated on a scale of 0 (not at all) to 3 (nearly every day) to represent how frequently the symptoms are experienced over the previous two weeks. A total score is calculated by summing the scores for each item, providing a severity score between 0 and 27. Higher scores represent more severe depression, and scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe and severe depression, respectively.
Change in Anxiety | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  General Anxiety Disorder- 7 (GAD-7) (Spitzer et al., 2006) will be used to assess the severity of anxiety. The GAD-7 includes 7 items that represent the DSM-IV (APA) clinical criteria. The items, such as "becoming easily annoyed or irritable", are scored on a scale between 0 (not at all) to 3 (nearly every day) to represent how frequently the symptoms are experienced over the previous two weeks. A total score between 0 - 21 is calculated by summing each individual item's rating. Higher scores represent more severe anxiety, and scores of 5, 10 and 15 are the cut-off points for mild, moderate and severe anxiety, respectively.
Change in Stress | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The Perceived Stress Scale (PSS, Cohen et al., 1983) will be used to measure participant's perception of stress. The 10-item self-report questionnaire includes four positively worded items and six negatively worded items that are rated on how frequently (never [0] - very often [4]) respondents perceive their lives as unpredictable, uncontrollable or overwhelming. Positively worded items are reverse scored, and each item response is summed to provide a total score of between 0 - 40 whereby higher scores equal higher perceived stress.
ADHD severity | Baseline.
  The Adult ADHD Self-report Scale (ASRS; Kessler, 2010) will be used as a screening tool to assess the frequency of ADHD symptoms and as a measuring tool to assess any changes in ADHD symptomatology over time. The measure was created in association with the World Health Organisation (WHO) and is based on the clinical criteria presented in the DSM-IV (APA, 2013). Part A is a 6-item questionnaire that assesses the frequency to which ADHD symptoms are present on a 5-point Likert Scale (Never - Always). It is recommended that individuals who report "sometimes", "often" or "very often" to the first three questions, or "often", "very often" to the final three questions four or more items, have symptoms highly consistent with ADHD.
Changes in self-criticism | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The Self-Critical Rumination Scale (SCRS, Smart et al., 2016) is a 10-item self-report questionnaire which measures the frequency of self-criticism on a 4-point scale from not at all (0) to very well (3). Self-criticism in this measure is conceptualised as a form of negative thinking that focuses on devaluing oneself. A total score is obtained by summing item responses, whereby higher scores equal greater self-criticism. Scores can range between 0 - 30.

SECONDARY OUTCOMES:
Fear of compassion | Baseline
  The Fears of Compassion for Self (FOC-FS) (Gilbert et al., 2011) subscale will measure the level of resistance respondents have in projecting compassion towards the self. The measure includes 15 items (e.g., "Getting on in life is about being tough rather than compassionate") that are rated on a scale between 0 (don't agree at all) ¬- 4 (completely agree). Item responses are summed to give a total score between 0 and 60 whereby higher scores indicate a greater fear of compassion towards the self.
Acceptability of the Intervention | Immediately following intervention end
  Acceptability of the intervention at post-intervention will be assessed following Sekhon et al.'s (2017) Theoretical Framework of Acceptability (TFA). A visual analogue rating scale will be used to measure: (1) affective attitude - how do you feel about the intervention?; (2) burden - how satisfied were you with the amount of time/effort the intervention required?; (3) ethicality - how well do you feel the intervention fits with your value system?; (4) self-efficacy - how confident are you that you could perform the intervention tasks?; (5) opportunity costs - to what extent did you have to give up something to take part in the intervention?; (6) perceived effectiveness - how confident are you that this intervention will improve your well-being?; (7) intervention coherence will be measured through a basic definitions quiz of self-compassion principles.
Change in daily Mood | Prior to each intervention session
  Mood will be measured daily using two affective sliders that rate level of alertness and level of happiness/pleasure on a 10-point scale. The two item responses are added together to give an overall score of mood between 0 and 20, whereby higher scores equal a more positive mood.
Change in ADHD trait severity | Baseline. Immediately following intervention end point. One month (4 weeks) following intervention end point.
  The Adult ADHD Self-report Scale (ASRS; Kessler, 2010) will be used as a measuring tool to assess any changes in ADHD symptomatology over time. The measure was created in association with the World Health Organisation (WHO) and is based on the clinical criteria presented in the DSM-IV (APA, 2013). It consists of 18 items that question the frequency of ADHD symptoms from "never" to "very often" (0 - 4) over the previous 6 months. Part A consists of 6-items that are most predictive of the disorder. Part B includes an additional 12 items which act as additional cues to participants symptoms. A total score can be obtained by summing the scores. A higher total score would represent a more frequent display of ADHD symptoms, and scores can range between 0 - 72.
Perfectionism | Baseline.
  Hewitt & Flett Multidimensional Perfectionism Scale (MPS-HW) Short form (2008), is a 15 item self-report questionnaire. Items are rated on a scale between 1-7 (Strongly disagree - strongly disagree), and is scored by summing responses to items. Higher scores indicate higher levels of perfectionism. Scores can range between 15 and 105.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All collected information will be anonymised and shared as part of open science protocol. Consent to share data will be obtained from participants prior to data collection.
Supporting Information: Analytic Code
Time Frame: When study results are accepted for publication.

REFERENCES:
- See also: self-compassion website where intervention exercises are found. — https://self-compassion.org/